CLINICAL TRIAL: NCT06759480
Title: Comparison Between Laparoscopic Radical Hysterectomy Based on Space Anatomy and Abdominal Radical Hysterectomy for Stage IB3 and IIA2 Cervical Cancer: a Multicenter Retrospective Cohort Study
Brief Title: Study of Laparoscopic Radical Hysterectomy Based on Space Anatomy in Patients With IB3 and IIA2 Cervical Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: International Peace Maternity and Child Health Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GKLW-A-2024-111-01
Record Dates: First submitted 2024-12-28; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Locally Advanced Cervical Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LRH group: In this group, patients received a modified laparoscopic radical hysterectomy(LRH) based on space antomy.
  Interventions: Procedure: Laparoscopic radical hysterectomy based on space anatomy
- ARH group: In this group, patients received a traditional abdominal radical hysterectomy(ARH). ARH group is defined as a control group.
  Interventions: Procedure: Abdominal radical hysterectomy

INTERVENTIONS:
Procedure: Laparoscopic radical hysterectomy based on space anatomy — This is a modified laparoscopic radical hysterectomy based on space anatomy. By identifying the vesicouterine ligament and four associated special spaces, the ureter can be completely liberated from the external aspect of the uterus. This skill not only reduces rate of surgical complications but also facilitates optimal tumor resection.
  Groups: LRH group
Procedure: Abdominal radical hysterectomy — This producre is a classic and traditional radical hysterectomy.
  Groups: ARH group

SUMMARY:
Radical hysterectomy is an effect treatment for FIGO IB3 and IIA2 cervical cancer patients who refuse to receive radical concurrent chemoradiotherapy. However, due to the large tumor size, both patients and surgeons encountered the risk of substantial bleeding, urinary tract damage, and unsatisfactory resection during surgery. Therefore, the exploration of effective and safe surgical treatments is crucial in enhancing the quality of life and prognosis for patients. Laparoscopic radical hysterectomy (LRH) offers the advantages of reduced bleeding and accelerated recovery, thereby minimizing patient discomfort and enhancing their quality of life. However, the prognosis of patients who received LRH or traditional abdominal radical hysterectomy (ARH) remains controversial. We proposed a modified LRH skill based on new space anatomy concept. In our previous single-center study, the result demonstrates that LRH based on space anatomy leads to less intraoperative blood loss and decreased ureteral injury rate compared with traditional skill. The benefits of this new method for patient survival remain uncertain. In this multicenter retrospective study, we aim to assess clinical prognosis and safety of this new LRH compared with traditional abdominal radical hysterectomy (ARH) in FIGO IB3 and IIA2 cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 20 to 70 years
2. Preoperative clinical diagnosis was FIGO 2018 stage IB3 or IIA2 cervical cancer;
3. Patients who received standard Querleu-Morrow type C radical hysterectomy (including ARH or LRH based on space anatomy) and pelvic lymphadenectomy;
4. no preoperative suspected lymph nodes metastasis, parametrial involvement or lower 1/3 vagina involvement.

Exclusion Criteria:

1. patients who had active double cancer or uncontrolled serious concurrent disease that might compromise prognosis;
2. pregnancy;
3. incomplete radical surgery;
4. follow-up time less than 6 months or lost to follow-up

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who clinically diagnosed with IB3 and IIA2 cervical cancer are retrospectively collected from electronic medical records of four tertiary medical center from January 2012 to January 2022
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-12-27 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  The time from end of surgery to death from any cause.
Progression-free survival | 5 years
  The time from end of surgery to either the first documented disease progression or death from any cause.

SECONDARY OUTCOMES:
Surgery complication rate | Intraoperative or within 2 weeks after surgery
  Including the rates of ureter or bladder injury, colon injury, deep vein thrombosis event and infection.
Intraoperative blood loss | Intraoperative blood loss

IPD SHARING:
Plan to Share IPD: Undecided